CLINICAL TRIAL: NCT02639754
Title: Community Intervention for HIV Testing & Care Linkage Among Young MSM in Bulgaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRO00024824; R01HD085833 (NIH)
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social Network Leader Endorsement (Experimental): Leaders of social networks randomized to this arm will be trained to endorse frequent HIV testing, compliance with medical guidelines, and effective ways to communicate these concepts to social network members.
  Interventions: Behavioral: Social Network Leader Endorsement
- Routine Counseling (Active Comparator): Members of social networks randomized to this arm will receive HIV counseling at baseline sessions.
  Interventions: Behavioral: HIV Counseling

INTERVENTIONS:
Behavioral: Social Network Leader Endorsement — Leaders of social networks will attend a multi-session intervention during which they will be trained to deliver messages endorsing frequent HIV testing, compliance with medical guidelines, and adherence to medical treatment regimens to friends. Additionally, these leaders will be trained on how to deliver effective messages.
  Arms: Social Network Leader Endorsement
Behavioral: HIV Counseling — At the baseline session, participants in this condition will receive counseling about the benefits and availability of HIV care and the importance of frequent HIV testing.
  Arms: Routine Counseling

SUMMARY:
Young men who have sex with men (MSM) in low- and middle-income countries often do not seek out HIV testing, are unaware of their HIV-positive status, and do not receive early medical care, compromising their health and contributing to downstream disease incidence. This situation is of great concern in post-socialist countries of Eastern Europe, where stigma about HIV/AIDS and same-sex behavior are great, HIV epidemics are still increasing, and the health needs of young MSM are rarely acknowledged or addressed. The planned research will be conducted in Sofia, Bulgaria, where MSM account for nearly half of HIV infections. The study will be conducted in two phases.

DETAILED DESCRIPTION:
In an initial qualitative phase, the investigators will conduct in-depth interviews with MSM ages 16 to 20 and other key informants to gain an understanding of factors related to HIV testing. The project's second phase is a trial of a network intervention to increase regular HIV testing and care linkage among young MSM. The investigators' prior studies in Bulgaria have shown that young MSM are clustered with other young MSM in social networks. The intervention trial will recruit 54 small social networks of MSM, each consisting of a young MSM "seed" between age 16 and 20 and also all close MSM friends surrounding the seed. All participants will complete baseline measures assessing recent HIV testing practices and testing history; attitudes, intentions, perceived norms, barriers, and understanding about HIV testing and medical care; sexual risk practices; and substance use. All participants will receive HIV risk reduction counseling. Networks will then be randomized to comparison and intervention conditions. Influence leaders of each experimental condition network will be identified, and network leaders will together attend a 5-session intervention, which will train, guide, and engage leaders to deliver theory-based, personally-tailored advice and counseling to their network members to correct misconceptions about HIV testing and care; strengthen friends' norms, attitudes, intentions, and perceived benefits of regular testing; and address barriers to testing. All members of intervention and comparison condition networks will be re-assessed at 6- and 12-month followup to determine the intervention's effects on HIV testing, regular testing, and testing- and care-related scale measures. Participants diagnosed with HIV infection at any point will be linked to medical care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must identify as male at birth;
* Individuals must report having sex with other males;
* Individuals will be between the ages of 16 and 20;
* Individuals must live in the greater Sofia metropolitan area;
* Individuals must be able to provide written informed consent.

Exclusion Criteria:

* Individuals who do not report they were male at birth;
* Individuals who do not report having sex with other males;
* Individuals younger than 16 or older than 20;
* Individuals who reside outside of the greater Sofia metropolitan area;
* Individuals who are unable to provide written informed consent.

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Actual)
Dates: Start 2015-12; Primary Completion 2020-11 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of HIV Testing | 6 months; 12 months
  Change in the number of HIV tests completed within the 6 months prior to baseline will be compared with the number of HIV tests completed 0-6 months post-intervention and 7-12 months post-intervention

SECONDARY OUTCOMES:
Change in Medical Appointment Keeping | 6 months; 12 months
  Changes in the number of medical appointments scheduled and kept relative to baseline will be compared at 6 and 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Health and Social Development Foundation, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No